CLINICAL TRIAL: NCT03371810
Title: Pilot Randomized-controlled Phase-IIa Trial on the Prevention of Comorbid Depression and Obesity in Attention-deficit/ Hyperactivity Disorder
Brief Title: Prevention of Comorbid Depression and Obesity in Attention-deficit/ Hyperactivity Disorder
Acronym: PROUD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Heidelberg University (Other); Radboud University Medical Center (Other); Hospital Vall d'Hebron (Other); King's College London (Other)
Responsible Party: Principal Investigator, Christine M. Freitag, Prof. Dr., Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CoCA-PROUD
Record Dates: First submitted 2017-03-03; First posted 2017-12-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Attention-Deficit / Hyperactivity Disorder; Depression; Obesity
Keywords: attention-deficit / hyperactivity disorder; depression; obesity; prevention; bright light therapy; exercise; mobile healthy system
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression; Obesity; Motor Activity | interventions — Ultraviolet Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, observer-blinded, controlled, multi-centre, pilot phase-IIa parallel-group design with three arms (two treatment groups and one control group); three trial phases: baseline assessment, 10 weeks of treatment versus treatment as usual; 12 weeks post-treatment observation period.
Who Masked: Outcomes Assessor
Masking Description: Observer-blinded assessment of the primary outcome measure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright light therapy (Experimental): Mobile therapeutic light (10.000 LUX), daily (except Sunday) for 30 min in the morning or evening for 10 weeks in total.
  Additional treatment as usual comprising pharmacotherapy, group based or individual cognitive behavioural therapy (not including elements of bright light therapy or exercise) is allowed.
  Interventions: Behavioral: Bright light therapy
- Physical exercise (Experimental): Aerobic exercise of moderate-to-vigorous intensity three days a week plus muscle-strengthening exercises two days a week during 10 weeks in total.
  Additional treatment as usual comprising pharmacotherapy, group based or individual cognitive behavioural therapy (not including elements of bright light therapy or exercise) is allowed.
  Interventions: Behavioral: Physical exercise
- Treatment as usual (No Intervention): Stable treatment as usual comprising pharmacotherapy, group based or individual cognitive behavioural therapy (not including elements of bright light therapy or exercise).

INTERVENTIONS:
Behavioral: Bright light therapy — Mobile therapeutic light (10.000 LUX, white light without UV light), daily (except Sunday) for 30 min in the morning or evening for 10 weeks in total at home provided by a bright light therapy device (Philips EnergyLight HF 3419). Monitoring and feedback will be realized with the m-Health system comprising of a smartphone equipped with the m-Health App, and an activity sensor equipped with a light sensor to monitor the light exposure of the participant.
  Other Names: Device: smartphone with m-Health app; Device: Philips EnergyLight HF 3419
  Arms: Bright light therapy
Behavioral: Physical exercise — During 10 weeks participants perform three days of aerobic activities proposed and in two of these days also do muscle-strengthening exercise. Specifically, a training day consists of: (i) a 5-min warm-up period, (ii) a 10-35 min of muscle-strength training on two of the three days, (iii) a 20-40 min of aerobic training, (iii), and a 5-min of flexibility/stretching cool-down. During the course of the 10 weeks, the duration and intensity of the exercises will increase gradually.
  Instruction, monitoring, and feedback will be realised by the m-Health system including a smartphone equipped with the m-Health app and Secure Digital Memory cards to store the exercise videos as well as an activity sensor equipped with a mobile sensor for the acquisition of physical activity.
  Other Names: Device: smartphone with m-Health app
  Arms: Physical exercise

SUMMARY:
Depression and obesity are very common among adolescents and young adults with attention-deficit/ hyperactivity disorder (ADHD). However, intervention programmes to prevent these comorbid disorders rarely exist. In a pilot randomized-controlled study we test two newly developed intervention programmes that do not involve medication: bright light therapy and physical exercise. Both interventions will be supported by a mobile Health application to monitor and feedback intervention success and booster patients' motivation.

DETAILED DESCRIPTION:
The risk for comorbid major depressive disorder and obesity is increased in adolescents and adults with attention-deficit/ hyperactivity disorder (ADHD), and adolescent ADHD predicts adults major depressive disorder and obesity. Nonpharmacological interventions to prevent these comorbidities are urgently needed. Bright light therapy (BLT) improves day-night rhythm and is an established therapy for major depression in adolescents and adults. Exercise prevents and reduces obesity in adolescents and adults and also improves depressive symptoms. Interestingly, a reinforcement-based intervention using a mobile health app (m-Health) resulted in improved effects on weightloss in obesity. The aim of the current pilot randomized-controlled phase-IIa study is to establish feasibility and effect sizes of two kinds of interventions, BLT and exercise, in combination with m-Health based monitoring and reinforcement in adolescents and young adults aged 14 to 45 years old with ADHD, targeting the prevention of depressive symptoms and obesity. In addition, immediate and long-term treatment effects on ADHD specific psychopathology, health related quality of life, fitness and body related measures, neurocognitive functions and chronotype are explored. Furthermore, saliva samples are taken in a subgroup of adult patients to explore the effects of BLT and exercise on concentrations of hormones. This subgroup of adult patients will also participate in an additional neuroimaging study of the reward system in order to explore intervention effects on striatal reward reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria
* Stable treatment as usual comprising pharmacotherapy, group based or individual cognitive behavioural therapy (not including elements of bright light therapy or exercise)

Exclusion Criteria:

* Intelligence Quotient (IQ) below 75
* Any severe (comorbid) psychiatric disorder with necessary additional psychopharmaco or daycare/ inpatient therapy beyond treatment as usual
* Severe medical/ neurological condition not allowing bright light therapy or exercise
* History of epilepsy
* Use of antipsychotics, antiepileptic or photosensitising medication
* Substance abuse/ dependency

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in clinician-rated depressive symptoms (observer-blinded assessment) | baseline, end of intervention (10 weeks after baseline)
  Inventory of Depressive Symptomatology (clinician-rated)

SECONDARY OUTCOMES:
Change from baseline in clinician-rated depressive symptoms (observer-blinded assessment) | baseline, follow up (22 weeks after baseline)
  Inventory of Depressive Symptomatology (clinician-rated)
Change from baseline in clinician-rated ADHD symptoms | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  ADHD Rating Scales for adults and children
Change from baseline in self-reported severity of depressive symptoms | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Beck Depression Inventory II
Change from baseline in self-reported health status | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Health Questionnaire EQ-5D-3L
Change from baseline in self-reported health related quality of life | baseline, end of intervention (10 weeks after baseline)
  Short Form Health Questionnaire General Health Questionnaire
Change from baseline in self-reported general health status | baseline, end of intervention (10 weeks after baseline)
  General Health Questionnaire General Health Questionnaire
Change from baseline in self-reported emotional and behavioural problems in adolescents | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Youth self-report
Change from baseline in self-reported emotional and behavioural problems in adults | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Adult self-report
Change from baseline in circadian rhythm | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Munich Chronotype Questionnaire
Change from baseline in cognitive emotion regulation | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Cognitive Emotion Regulation Questionnaire
Change from baseline in neurocognitive functions: verbal memory | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Rey Auditory Verbal Learning Test
Change from baseline in neurocognitive functions: Digit span | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Digit span
Change from baseline in self-reported physical fitness | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  International Fitness Scale
Change from baseline in general muscular fitness | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  handgrip strength test
Change from baseline in muscular fitness | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  standing long jump test
Change from baseline in aerobic fitness | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  Chester step test
Change from baseline in body mass index | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  body mass index measured by clinician
Change from baseline in waist circumference | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  waist circumference measured by clinician
Change from baseline in waist-to-hip ratio | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  waist-to-hip ratio measured by clinician
Change from baseline in body fat percentage | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  based on skinfold thickness measurements using a skinfold caliper
Change from baseline in heart rate | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  heart rate measured by clinician
Change from baseline in blood pressure | baseline, end of intervention (10 weeks after baseline), follow-up (22 weeks after baseline)
  blood pressure measured by clinician
Change from baseline in number of steps | baseline, end of intervention (10 weeks after baseline)
  number of steps measured with the mobile Health app
Change from baseline in movement acceleration | baseline, end of intervention (10 weeks after baseline)
  movement acceleration measured with the mobile Health app
Change from baseline in sleep time | baseline, end of intervention (10 weeks after baseline)
  sleep time measured with the mobile Health app
Change from baseline in context parameters | baseline, end of intervention (10 weeks after baseline)
  context measured with the mobile Health
Change from baseline in mood regulation | baseline, end of intervention (10 weeks after baseline)
  mood regulation measured with the mobile Health app
Change from baseline in reward reactivity | baseline, end of intervention (10 weeks after baseline)
  reward reactivity measured with the mobile Health app
Change from baseline in stress reactivity | baseline, end of intervention (10 weeks after baseline)
  stress reactivity measured with the mobile Health app
Change from baseline in inattention | baseline, end of intervention (10 weeks after baseline)
  inattention measured with the mobile Health app
Change from baseline in melatonin concentration | baseline, end of intervention (10 weeks after baseline)
  Saliva sample will be taken to measure melatonin concentration
Change from baseline in cortisol concentration | baseline, end of intervention (10 weeks after baseline)
  Saliva sample will be taken to measure cortisol concentration
Change from baseline in leptin concentration | baseline, end of intervention (10 weeks after baseline)
  Saliva sample will be taken to measure leptin concentration
Change from baseline in ghrelin concentration | baseline, end of intervention (10 weeks after baseline)
  Saliva sample will be taken to measure ghrelin concentration
Change from baseline in neural activity associated with reward processing | baseline, end of intervention (10 weeks after baseline)
  Striatal functional magnetic resonance imaging signal related to reward processing

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Freitag, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital, Goethe University Frankfurt am Main
Locations (4):
- Goethe University Hospital Frankfurt, Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, and Department of Psychiatry, Psychosomatic Medicine and Psychotherapy, Frankfurt am Main, Germany
- Radboud University Medical Centre, Karakter Child and Adolescent Psychiatry, and Department of Psychiatry, Nijmegen, Netherlands
- Vall d'Hebron Research Institute, Group of Psychiatry, Mental Health and Addiction, Barcelona, Spain
- King's College London, Social, Genetic and Developmental Psychiatry Centre, Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mayer JS, Kohlhas L, Stermann J, Medda J, Brandt GA, Grimm O, Pawley AD, Asherson P, Sanchez JP, Richarte V, Bergsma D, Koch ED, Muntaner-Mas A, Ebner-Priemer UW, Kieser M, Retz W, Ortega FB, Colla M, Buitelaar JK, Kuntsi J, Ramos-Quiroga JA, Reif A, Freitag CM. Bright light therapy versus physical exercise to prevent co-occurring depression in adolescents and young adults with attention-deficit/hyperactivity disorder: a multicentre, three-arm, randomised controlled, pilot phase-IIa trial. Eur Arch Psychiatry Clin Neurosci. 2025 Apr;275(3):653-665. doi: 10.1007/s00406-024-01784-1. Epub 2024 Apr 16. PMID 38627266
- [Derived] Mayer JS, Hees K, Medda J, Grimm O, Asherson P, Bellina M, Colla M, Ibanez P, Koch E, Martinez-Nicolas A, Muntaner-Mas A, Rommel A, Rommelse N, de Ruiter S, Ebner-Priemer UW, Kieser M, Ortega FB, Thome J, Buitelaar JK, Kuntsi J, Ramos-Quiroga JA, Reif A, Freitag CM. Bright light therapy versus physical exercise to prevent co-morbid depression and obesity in adolescents and young adults with attention-deficit / hyperactivity disorder: study protocol for a randomized controlled trial. Trials. 2018 Feb 26;19(1):140. doi: 10.1186/s13063-017-2426-1. PMID 29482662
- See also: Homepage of the CoCA project (Comorbid Conditions of Attention-deficit / hyperactivity disorder).The PROUD study is work package 6 of the CoCA project. — http://coca-project.eu/coca-phase-iia-trial/study/